CLINICAL TRIAL: NCT04702126
Title: Smoking Effect on Lumbar Intervertebral Disc Degeneration
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, fatma esra bahadir ulger, Fatih Sultan Mehmet Training and Research Hospital, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRHU
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Intervertebral Disc Degeneration
Keywords: Intervertebral disc degeneration; Magnetic resonance imaging; Smoking; Passive smoker
MeSH Terms: conditions — Intervertebral Disc Degeneration; Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Besides normal aging, genetic and environmental factors are important potential determinants of lumbar disc degeneration. Smoking causes serious health problems, particularly lung and other cancers, heart disease and respiratory diseases, and is among the most common causes of death worldwide. Besides these commonly known diseases related to smoking numerous studies have shown that smoking has detrimental effects on the musculoskeletal system and worsens the prognosis and treatment of leukomotor diseases. In the literature there are studies examining the effect of smoking status on disc degeneration. The aim of the study was to investigate the effect of current, former and passive smoking status on degeneration of lumbar intervertebral discs.

DETAILED DESCRIPTION:
This retrospective study was performed by obtaining medical records of patients who underwent lumbar spinal MRI between September 2019 and February 2020. After the application of exclusion criteria 955 patients determined between the specified dates. These patients were called by phone to be questioned about their smoking status and whether they were working in heavy work and whether they were athletes. Heavy workers and athletes were also excluded from the study and a total of 360 patients whose smoking status information could be obtained were included in the study.The patients were grouped according to their smoking status as "current smoker", "former smoker", "non-smoker" and "passive smoker". The cumulative smoking dose for current and former smokers was calculated in terms of pack-years and categorized further into two subgroups: smoked ≤9 pack-years or >9 pack-years. The number of pack-years was calculated by dividing the number of cigarettes consumed per day by 20 and multiplying by the years that the patient had smoked. Age, gender, weight, and height were recorded, and body mass index (BMI) was calculated as weight/(height)2. Lumbar spinal MRI was performed using a 1.5 Tesla imaging system (General Electric Healthcare, Milwaukee, WI), using the following settings: amplitude: 44 mT/m; slew rate gradient configuration: 200 T/m/s. MRI images were evaluated using a GE Advantage Workstation (GE Healthcare, Buc, France) and Volume Share software v.7.0. The lumbar lordosis angle was measured and the lumbar intervertebral discs were evaluated by Pfirrmann disc degeneration grading system using sagittal T2-weighted MR images (TR/TE: 2500/85 ms, matrix: 320x224, slice thickness: 4 mm, FOV: 32) (23). The degree of degeneration was classified into five grades with Grades IV and V considered as "severe disc degeneration". Radiologist reviewing the MRI studies was blinded to the smoking status of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent lumbar spinal MRI between September 2019 and February 2020.

Exclusion Criteria:

* a history of spinal surgery or instrumentation, spinal fracture, trauma, congenital or acquired spinal deformity tumor or infection,
* heavy physical workers,
* athletes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lumbar spinal MRI between September 2019 and February 2020 and questioned for smoking status.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of current, former and passive smoking status on degeneration of lumbar intervertebral discs. | 3 months
  The lumbar intervertebral discs of patients were evaluated by Pfirrmann disc degeneration grading system using sagittal T2-weighted MR images. The degree of degeneration was classified into five grades with Grades IV and V considered as "severe disc degeneration". Severe disc degeneration was identified between the current, former, passive and non-smoker groups. The relationship between smoking status groups and severe disc degeneration was examined.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Esra Bahadir Ülger, M.D., Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)